CLINICAL TRIAL: NCT06972667
Title: Interventions to Decrease Cancer Information Avoidance
Brief Title: Interventions to Decrease Health Information Avoidance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather Orom, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00009059; R01CA276430 (NIH)
Record Dates: First submitted 2025-05-03; First posted 2025-05-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Health Information Avoidance
Keywords: colorectal cancer screening; information avoidance; RCT; screening intentions; video

STUDY DESIGN:
Intervention Model Description: The study will be a randomized controlled trial. Participants (N=1,500), half of whom will be selected because they tend to avoid colorectal cancer information, will be randomized to treatment groups using a stratified permuted block randomization scheme to ensure equal proportion of avoiders across videos.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video to promote colonoscopy (Experimental): Participants will view a brief video promoting colonoscopy with self-efficacy enhancement, humor and calm affect induction
  Interventions: Other: Video to promote colonoscopy
- Video to promote screening for colorectal cancer with home tests (Experimental): Participants will view a brief video promoting colorectal cancer home testing with self-efficacy enhancement, humor and calm affect induction
  Interventions: Other: Video to promote screening for colorectal cancer with home tests
- Attentional control video (No Intervention): The attentional control video will be about food safety and will be the same length and include the same actors and music.

INTERVENTIONS:
Other: Video to promote colonoscopy — This video contains elements designed to engage and persuade people who tend to avoid colorectal cancer information to have a colonoscopy. Psychological elements include self-efficacy boosting, humor, and calming affect induction.
  Arms: Video to promote colonoscopy
Other: Video to promote screening for colorectal cancer with home tests — This video contains elements designed to engage and persuade people who tend to avoid colorectal cancer information to screen for colorectal cancer with a home test. Psychological elements include self-efficacy boosting, humor, and calming affect induction.
  Arms: Video to promote screening for colorectal cancer with home tests

SUMMARY:
Health information avoidance is an overlooked threat to the reach and effectiveness of health communication. To fully realize the benefits of our sizeable investments in health messaging, it is necessary to identify strategies for reducing health information avoidance. The researchers will test a video-based strategy for promoting colorectal cancer screening designed to reduce defensive colorectal cancer information avoidance and increase message reach by increasing engagement among those who would otherwise avoid the message. The researchers will conduct a randomized controlled trial (RCT) comparing the effects of the intervention video to an attentional control video on colorectal cancer screening intentions and uptake.

DETAILED DESCRIPTION:
The study will test the efficacy and mediating mechanisms of brief video interventions including elements demonstrated to be effective in reducing health information avoidance (self-efficacy boosting, humor, calm affect induction). It is expected that the videos to benefit people who typically avoid health information yet still be beneficial for people who do not avoid health information, thus being suitable for dissemination to general audiences. It is hypothesized that the interventions will strengthen intentions to be screened, increase colorectal cancer risk information seeking and increase screening.

Following recommended practices, the two intervention arms and the control arm will include multiple versions of the videos to control for actor effects. All intervention videos operationalize the same psychological mechanisms but are delivered by 4 different actors and promote either colonoscopy or stool tests. The 8 parallel intervention and 4 control videos will be treated as random effects.

The intervention videos will be tested in members of the Ipsos panel who are not adherent to colorectal cancer screening guidelines, half of whom will be selected because they tend to avoid colorectal cancer information. Effects of the intervention videos will be compared to those of an attentional control video about food safety.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 45 and 75 years
* never diagnosed with colorectal cancer
* non-adherent to colorectal cancer screening guidelines
* half will have a score at or greater than the mid-point on the colorectal cancer information avoidance scale (≥2.5) on the pre-screening survey such that half of the sample are people who tend to avoid colorectal cancer information

Exclusion Criteria:

* not between the ages of 45 and 75 years
* have been diagnosed with colorectal cancer
* adherent to colorectal cancer screening guidelines

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Strength of screening intentions | Day 1
  Participants will rate their intention to be screened with the item, "I intend to get checked for colon cancer within the next 6 months" on a scale from 1 to 4 with 4 being stronger intentions.
Strength of intentions to talk to a health care provider about being screened for colorectal cancer | Day 1
  This outcome will be assessed with the item, "I will talk to a health care provider about getting checked for colon cancer within the next 6 months".
Proportion of participants who seek personal risk information | Day 1
  Participants will be asked whether they want to be redirected at the end of the study to complete the online Siteman Cancer Center colorectal cancer risk calculator.
Proportion of participants screened for colorectal cancer after 9 months | At least 9 months after start of study
  The researchers will assess whether participants have been screened for colorectal cancer in the 9 months since participating in the intervention phase of the study.

SECONDARY OUTCOMES:
Self-efficacy for colorectal cancer screening | Day 1
  Sel-efficacy will be assessed with 2 items with which participants rate their confidence in arranging to get screened and completing a screening test on a scale ranging from 0 to 10, with 10 indicating greater self-efficacy.
Positive and negative affect | Day 1
  Positive and negative affect will be assessed with the Positive and Negative Affect Schedule Short Form (PANAS-SF). Scores range from 1 to 5, with higher scores indicating more of a given affect.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Orom Associate Professor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All non-identifying study data will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: IPD will be available once results are published. There will be no end date.
Access Criteria: Anyone will be able to access the IDP through OSF.
URL: https://osf.io/

DOCUMENTS (1):
  • Informed Consent Form (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT06972667/ICF_000.pdf